CLINICAL TRIAL: NCT04834817
Title: The Effect of Combined Red and Near Infrared Light-emitting Diode (LED) Therapy on Tissue Regeneration Post Laser Treatment
Brief Title: Effect of Combined Red and Near Infrared Light-emitting Diode (LED) Therapy on Tissue Regeneration Post Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: BioPhotas (Industry)
Responsible Party: Principal Investigator, Kristen Kelly, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20216401
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Wound Heal

STUDY DESIGN:
Intervention Model Description: This is a split-person study design where each participant has one arm with the intervention and the other arm that is control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LED treatment (Experimental): LED treatment with Celluma POD device after laser test area
  Interventions: Device: Celluma POD
- Control (No Intervention): No treatment after laser test area

INTERVENTIONS:
Device: Celluma POD — A blue and near infrared handheld LED device
  Arms: LED treatment

SUMMARY:
The purpose of this study is to evaluate the effect of light therapy on wound healing after laser treatment.

DETAILED DESCRIPTION:
This study sets out to evaluate the effect of a combination of near infrared (830 nm) red (633 nm) and blue (465nm) light-emitting diode (LED) therapy on wound healing after laser application.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older with no active cutaneous disease on bilateral ventral biceps, close to the axilla.

Subjects shall have given written informed consent for both the LED therapy and for clinical photography.

Exclusion Criteria:

Patients will be excluded if any of the exclusion criteria applies

* Subjects refuse to give informed consent for either the phototherapy or the clinical photography.
* Subjects have previous photosensitivity problems (solar urticaria, etc.).
* Subjects are taking any systemic drug or applying any topical drug with known photosensitizing properties.
* Subjects taking any systemic drug with known immunosuppressant properties.
* Subjects applying any medications to the research site (inner biceps, close to the axilla).
* Subjects have medical or psychosocial conditions associated with a risk of poor protocol compliance.
* Subjects are smokers or have smoked within the last 30 days prior to the trial.
* Subjects have epilepsy or a history of seizures
* Subjects currently taking cortisone injections or any other kind of steroid injections(s)
* Subjects with known cancer tumor in the treatment area or metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Beckman Laser Institute and Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: wound area
Period: Overall Study
Arm/Group | LED Treatment | Control
Started | 25; 25 wound area | 25; 25 wound area
Completed | 25; 25 wound area | 25; 25 wound area
Not Completed | 0; 0 wound area | 0; 0 wound area

BASELINE CHARACTERISTICS:
Population: 32 subjects were screened and consented. 7 subjects were unable to participate due to scheduling difficulties. They never participated in any study procedures. 25 subjects participated in the study as both experimental and control groups.
Units Other Than Participants: wound area
Groups:
- Total: Total of all reporting groups
Arm/Group | LED Treatment | Control | Total
Number analyzed (Participants) | 25 | 25 | 25
Number analyzed (wound area) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: Age] | 37 [19 to 65] | 37 [19 to 65] | 37 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Units; unit: wound area]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Race (NIH/OMB) [Count of Units; unit: wound area]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Days to Healing
Description: The primary endpoint of this study is time and days to complete healing of the treatment sites. Clinical grading shall be by blinded assessment.
Time Frame: Assessed from Day 0 to Day 55, up to 56 days
Measure: Number; unit: participants
Arm/Group | LED Treatment | Control
Number analyzed (Participants) | 25 | 25
participants
  Erythema healed by day 27 | 24 | 24
  Erythema resolved by day 34 | 1 | 0
  Erythema resolved by day 55 | 0 | 1
  Edema resolved by day 4 | 25 | 24
  Edema resolved by day 27 | 0 | 1
  Crusting resolved by day 13 | 22 | 22
  Crusting resolved by day 27 | 3 | 3

2. Secondary Outcome: Pain Level
Description: A secondary outcome measure will be post-treatment pain on a 11-point Lickert scale from 0-10. Higher scores mean a worse outcome.
Time Frame: Assessed from Day 0 to Day 13, up to 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | LED Treatment | Control
Number analyzed (Participants) | 25 | 25
Participants
  Pain/discomfort-free on day 4 | 23 | 23
  Pain/discomfort-free on day 6 | 2 | 2
  Reported itch on days 9 and 13, resolved by day 13 | 3 | 0

ADVERSE EVENTS:
Time Frame: 55 days post-treatment
Arm/Group | LED Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04834817/Prot_SAP_000.pdf